CLINICAL TRIAL: NCT02193971
Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Diseases Trial - Comparison of REDUCTION of PrasugrEl Dose & POLYmer TECHnology in ACS Patients (HOST REDUCE POLYTECH RCT Trial) Comparison of the Efficacy and Safety of Biostable Polymer DES (Promus PremierTM, Xience Alpine®, and Resolute Onyx®) With Biodegradable Polymer DES (Biomatrix®, Biomatrix Flex®, Nobori®, Ultimaster®,Synergy®, and Orsiro®)and Conventional Dose Prasugrel Therapy With Reduced Dose Prasugrel Therapy in Acute Coronary Syndrome Patients Treated With Percutaneous Coronary Intervention
Brief Title: Harmonizing Optimal Strategy for Treatment of Coronary Artery Diseases Trial - Comparison of REDUCTION of PrasugrEl Dose & POLYmer TECHnology in ACS Patients (HOST REDUCE POLYTECH RCT Trial)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Boston Scientific Korea Co. Ltd (Industry); Dio (Industry); Terumo Corporation (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOST REDUCE POLYTECH RCT
Record Dates: First submitted 2014-07-13; First posted 2014-07-18 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Drug eluting stent; Everolimus; Prasugrel
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BS-DES with prasugrel 10mg daily (Active Comparator): BS-DES with prasugrel 10mg daily
  Interventions: Device: BS-DES (Biostable polymer drug-eluting stent)
- BS-DES with prasugrel 5mg daily (Active Comparator): BS-DES with prasugrel 5mg daily
  Interventions: Device: BS-DES (Biostable polymer drug-eluting stent); Drug: Prasugrel 5mg
- BD-DES with prasugrel 10mg daily (Experimental): BD-DES with prasugrel 10mg daily
  Interventions: Device: BD-DES (Biodegradable polymer drug-eluting stent)
- BD-DES with prasugrel 5mg daily (Experimental): BD-DES with prasugrel 5mg daily
  Interventions: Device: BD-DES (Biodegradable polymer drug-eluting stent); Drug: Prasugrel 5mg

INTERVENTIONS:
Device: BS-DES (Biostable polymer drug-eluting stent)
  Other Names: Promus Premier; Xience Alpine; Resolute Onyx
  Arms: BS-DES with prasugrel 10mg daily; BS-DES with prasugrel 5mg daily
Device: BD-DES (Biodegradable polymer drug-eluting stent)
  Other Names: Biomatrix; Biomatrix Flex; Nobori; Ultimaster; Synergy; Orsiro
  Arms: BD-DES with prasugrel 10mg daily; BD-DES with prasugrel 5mg daily
Drug: Prasugrel 5mg — Use prasugrel 5mg daily for maintaning dose
  Other Names: Prasugrel
  Arms: BD-DES with prasugrel 5mg daily; BS-DES with prasugrel 5mg daily

SUMMARY:
* Study objectives

  1. To compare the safety and long-term efficacy of coronary stenting with biostable polymer drug-eluting stent (Promus PremierTM, Xience Alpine®, Resolute Onyx®) with biodegradable polymer drug-eluting stent (Biomatrix®, Biomatrix Flex®, Nobori®, Ultimaster®, Synergy ® and Orsiro®) in patients with acute coronary syndrome
  2. To compare the efficacy and safety of 5 mg prasugrel maintenance therapy compared with 10 mg prasugrel maintenance therapy in patients with acute coronary syndrome undergoing percutaneous coronary intervention
* Study design :

Prospective, open-label, 2-by-2 multifactorial, randomized, multicenter trial to test the following in CHD patients

1. Non-inferiority of biostable polymer drug-eluting stent (Promus PremierTM, Xience Alpine®, Resolute Onyx®) compared with biodegradable polymer drug-eluting stent (Biomatrix®, Biomatrix Flex®, Nobori®, Ultimaster®, Synergy ® and Orsiro®) in terms of patient-oriented composite outcome
2. Non-inferiority of 5 mg compared to 10 mg dose of prasugrel maintenance in terms of major adverse cardiovascular events

DETAILED DESCRIPTION:
About 3400 patients derived from a population of Korean patients with acute coronary syndrome receiving percutaneous coronary intervention will be enrolled in the present trial.

All patients will receive a loading dose of aspirin (300 mg) and prasugrel (60 mg bolus) will be administered. Sixty-mg-loading dose of prasugrel will be given regardless of pretreated antiplatelet agents (clopidogrel, ticagrelor, or cilostazol). However, in patients who already loaded with other antiplatelet agents (clopidigrel, ticagrelor, or cilostazol), reduced dose (30mg) or omission of prasugrel loading is acceptable. Following angiography, patients with significant diameter stenosis >50% of coronary artery or graft vessel by visual estimation that have documented myocardial ischemia or symptoms of angina, and have lesions that are eligible for coronary intervention without any exclusion criteria, will be randomized 1:1 to either receive either BS-DES or BD-DES group.

At 1-month clinical follow-up, patients eligible for antiplatelet comparison will be additionally randomized 1:1 to either receive the reduce dose of prasugrel (5 mg daily) or conventional dose (10 mg daily). The exclusion criteria (age ≥75 years, body weight <60 kg, or history of TIA or stroke) is classified as observational cohort. Post-PCI, dual antiplatelet therapy is recommended for at least 1 year. Follow-up data will be collected until 3-year after index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Subject must have a culprit lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation
* Subject must have clinical diagnosis of acute coronary syndrome

Exclusion Criteria:

* Following patients will be enrolled in stent comparison, but excluded from antiplatelet comparison. They will be classified as observational cohort.
* Subjects ≥75 years
* Body weight <60 kg
* History of TIA or stroke
* The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Biolimus, Everolimus, Contrast media (Patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled.)
* Patients with active pathologic bleeding
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* Systemic (intravenous) Biolimus, or everolimus use within 12 months.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study.
* History of bleeding diathesis, known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3384 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-10 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Stent arm : patient-oriented composite outcome (POCO), defined as a composite of all death, myocardial infarction (MI) or repeat revascularization | 12months
Antiplatelet arm : major adverse cardiovascular event (MACE), defined as a composite of all death, MI, stent thrombosis, repeat revascularization, CVA, and BARC class ≥2 bleeding | 12months

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee KS, Park KH, Park KW, Rha SW, Hwang D, Kang J, Han JK, Yang HM, Kang HJ, Koo BK, Lee NH, Rhew JY, Chun KJ, Lim YH, Bong JM, Bae JW, Lee BK, Kim SY, Shin WY, Lim HS, Park K, Kim HS. Prasugrel dose de-escalation in diabetic patients with acute coronary syndrome receiving percutaneous coronary intervention: results from the HOST-REDUCE-POLYTECH-ACS trial. Eur Heart J Cardiovasc Pharmacother. 2023 Apr 10;9(3):262-270. doi: 10.1093/ehjcvp/pvad008. PMID 36715152
- [Derived] Hwang D, Lim YH, Park KW, Chun KJ, Han JK, Yang HM, Kang HJ, Koo BK, Kang J, Cho YK, Hong SJ, Kim S, Jo SH, Kim YH, Kim W, Lee SY, Kim YD, Oh SK, Lee JH, Kim HS; HOST-RP-ACS investigators. Prasugrel Dose De-escalation Therapy After Complex Percutaneous Coronary Intervention in Patients With Acute Coronary Syndrome: A Post Hoc Analysis From the HOST-REDUCE-POLYTECH-ACS Trial. JAMA Cardiol. 2022 Apr 1;7(4):418-426. doi: 10.1001/jamacardio.2022.0052. PMID 35262625
- [Derived] Kim HS, Kang J, Hwang D, Han JK, Yang HM, Kang HJ, Koo BK, Kim SY, Park KH, Rha SW, Shin WY, Lim HS, Park K, Park KW; HOST-REDUCE-POLYTECH-ACS Trial Investigators. Durable Polymer Versus Biodegradable Polymer Drug-Eluting Stents After Percutaneous Coronary Intervention in Patients with Acute Coronary Syndrome: The HOST-REDUCE-POLYTECH-ACS Trial. Circulation. 2021 Mar 16;143(11):1081-1091. doi: 10.1161/CIRCULATIONAHA.120.051700. Epub 2020 Nov 18. PMID 33205662
- [Derived] Kim HS, Kang J, Hwang D, Han JK, Yang HM, Kang HJ, Koo BK, Rhew JY, Chun KJ, Lim YH, Bong JM, Bae JW, Lee BK, Park KW; HOST-REDUCE-POLYTECH-ACS investigators. Prasugrel-based de-escalation of dual antiplatelet therapy after percutaneous coronary intervention in patients with acute coronary syndrome (HOST-REDUCE-POLYTECH-ACS): an open-label, multicentre, non-inferiority randomised trial. Lancet. 2020 Oct 10;396(10257):1079-1089. doi: 10.1016/S0140-6736(20)31791-8. Epub 2020 Aug 31. PMID 32882163
- [Derived] Lee JM, Jung JH, Park KW, Shin ES, Oh SK, Bae JW, Rhew JY, Lee N, Kim DB, Kim U, Han JK, Lee SE, Yang HM, Kang HJ, Koo BK, Kim S, Cho YK, Shin WY, Lim YH, Rha SW, Kim SY, Lee SY, Kim YD, Chae IH, Cha KS, Kim HS. Harmonizing Optimal Strategy for Treatment of coronary artery diseases--comparison of REDUCtion of prasugrEl dose or POLYmer TECHnology in ACS patients (HOST-REDUCE-POLYTECH-ACS RCT): study protocol for a randomized controlled trial. Trials. 2015 Sep 15;16:409. doi: 10.1186/s13063-015-0925-5. PMID 26374625